CLINICAL TRIAL: NCT04307459
Title: Acute Respiratory Failure and Continuous Positive Airway Pressure Therapy in Patients With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection: a Real Life Evaluation
Brief Title: Acute Respiratory Failure and COVID-19 in Real Life
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pierachille Santus, MD, PhD, Professor, Head of Respiratory Disease Unit H sacco, University of Milan
Other Study IDs: 17263/2020
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus Infections; Respiratory Failure; Ventilator Lung
Keywords: sars; acute respiratory failure; CPAP therapy; non invasive ventilation; gas exchange
MeSH Terms: conditions — Coronavirus Infections; Respiratory Insufficiency; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronavirus Infection: All patients admitted to the Respiratory Unit with SARS-CoV-2 infection and respiratory failure
  Interventions: Other: standard operating procedures

INTERVENTIONS:
Other: standard operating procedures — standard operating procedures represented by continuous positive airway pressure (CPAP) therapy or non invasive ventilation, pharmacological treatment as antiviral and antibiotic drugs, bronchodilators, xanthines, enteral nutrition, hydration.

SUMMARY:
In December 2019 a new kind of virus was identified in China as the responsible of severe acute respiratory syndrome (SARS) and interstitial pneumonia. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) quickly spread around the world and in February 2020 became a pandemia in Europe.

No pharmacological treatment is actually licensed for the SARS-CoV2 infection and at the current state of art there is a lack of data about the clinical management of the coronavirus 2019 disease (COVID-19).

The aim of this observational study is to collect the data and the outcomes of COVID-19 patients admitted in the H. Sacco Respiratory Unit treated according to the Standard Operating Procedures and the Good Clinical Practice.

DETAILED DESCRIPTION:
All consecutive adult COVID-19 patients admitted to our Respiratory Unit will be enrolled. All demographic, anthropometric, laboratory, radiological, clinical and microbiological data will be collected and analyzed according to the primary and secondary outcomes (see the dedicated section).

During the hospitalization, patients will be treated according to the standard operating procedure of our Respiratory Unit, such as arterial gas analysis, Rx, pharmacological treatment, ventilation. This study is purely observational and no randomization will be performed.

After discharge, patients a 7 days, 30 days and 6 months follow up will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients that can give written or oral informed consent
* patients with microbiological diagnosis (i.e. rhinopharyngeal swab) of SARS-CoV2 infection

Exclusion Criteria:

* severe cognitive impairment
* absolute contraindication to non invasive ventilation or cpap therapy
* rhinopharyngeal swab negative for SARS-CoV2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with SARS-CoV2 pulmonary disease admitted to the H. Sacco respiratory unit will be enrolled in the observational study (see exclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Real life data of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection | 1-6 months
  Data collection about the real life management of patients affected by SARS-CoV-2 infection with acute respiratory distress syndrome

SECONDARY OUTCOMES:
in-hospital mortality | 1 month
  How many patients died during the hospitalization
30 days mortality | 1 month
  How many patients died 30 days after the discharge
6 months mortality | 6 months
  How many patients died 6 months after the discharge
Intubation rate | 7 days
  How many patients were intubated during the hospitalization
Time to Intubation | 7 days
  How many days/hours from admittance to intubation
Time to ventilation | 7 days
  How many days/hours from admittance to the start of non invasive ventilation or CPAP therapy
Non invasive to Invasive time | 7 days
  How many days/hours from the start of non invasive ventilation or CPAP therapy to the intubation
Recovery rate | 1 month
  How many patients were healed from the infection and discharged
Recurrence rate | 1 month
  How many patients underwent re-infection after previous recovery from COVID19
Risk factor for COVID19 | retrospective
  Assessment of the risk factors for the infection and the admission to the hospital
Blood tests and outcome | 1 month
  What serological parameter could be used as predictor of good or negative prognosis.
Antiviral therapy | 1 month
  Impact of antiviral therapy on the clinical course of the disease
Coinfections | 1 month
  Assessment of bacterial, fungal or other coinfections rate
Radiological findings | 1 month
  Impact of radiological findings on the clinical course and the outcome
Ultrasound findings | 1 month
  Impact of ultrasound findings on the clinical course and the outcome
Myocardial injury | 1 month
  Assessment of the evidence of myocardial injury in covid19+ patients
Medical management | 1 month
  impact of standard therapeutic operating procedures (eg enteral nutrition, hydration, drugs) on the clinical course.

CONTACTS AND LOCATIONS:
Locations (1):
- Luigi Sacco University Hospital, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santus P, Radovanovic D, Saderi L, Marino P, Cogliati C, De Filippis G, Rizzi M, Franceschi E, Pini S, Giuliani F, Del Medico M, Nucera G, Valenti V, Tursi F, Sotgiu G. Severity of respiratory failure at admission and in-hospital mortality in patients with COVID-19: a prospective observational multicentre study. BMJ Open. 2020 Oct 10;10(10):e043651. doi: 10.1136/bmjopen-2020-043651. PMID 33040020